CLINICAL TRIAL: NCT02444702
Title: Clinical, Morphological and Functional Success Predictors Following Lumbar Spinal Surgery in Patients With Chronic Low Back Pain and Degenerative Disorders.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0006-15-MMC
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain
Keywords: spinal stenosis, clinical predictors rules, MRI, fusion, low back pain
MeSH Terms: conditions — Low Back Pain; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CLBP and degenerative lumbar spine: Participants with CLBP (>12 weeks) and degenerative changes of the lumbar spine confirmed by CT imaging who were recommended surgery and chose to undergo surgery will be recruited from the department of Orthopedic Surgery at the Meir Medical Center, Kfar-Saba, Israel. Included participants will be men or women, aged 40-80 years, of any race or ethnic background. Participants' diagnosis may include unstable degenerative spondylolisthesis, radicular pain, or documented stenosis with referred pain.

SUMMARY:
The long term goal of this project is dual fold. First, the investigators wish to derive, validate and then test the impact of a clinical prediction rule to determine which patients who suffer from CLBP with degenerative changes of the lumbar spine and referred pain to the legs are likely to require surgery and have successful outcomes in the long term. Second, the investigators would like to establish robust methodology and statistical analysis guidelines for creating clinical prediction rules in physical therapy research. This observational cohort project is a first step towards those goals. Here the investigators specifically aim to identify personal, behavioral, psychological, morphological, and physical factors that can predict the need for surgery as well as level of participation restriction in patients who suffer from CLBP with degenerative conditions of the lumbar spine and referred pain to the legs. The investigators will also explore which parameters can predict success after 1 month, 6 and 12 months in patients who underwent decompression/fusion surgery.

DETAILED DESCRIPTION:
A classification-based approach to identify specific characteristics of patients who seriously suffer from chronic low back pain (CLBP) with referred pain to the legs who are likely to respond to certain interventions has become a research priority in the medical milieu in general and in physical therapy in particularly.While several classifications have been developed to predict success following physical therapy interventions, some have methodological flaws and no clinical prediction rules have been created for patients with CLBP with degenerative changes of the lumbar spine and referred pain to the legs who are likely to require surgery and have successful outcome post-surgery. CLBP is multifactorial and morphological findings such as degenerative changes of the lumbar spine may not explain the phenomenon in full. The international classification of functioning, disability and health allows for a comprehensive description of the patient as a whole and can be used to classify patients according to their anatomy, pathology, impairments and capacity One-hundred and fifty patients who suffer from CLBP with degenerative conditions of the lumbar spine and referred pain to the legs and are candidates for lumbar decompression/fusion surgery will be recruited from a physician office at the Meir medical center, department of orthopaedic surgery, "Kfar-Saba", Israel. The structure and pathology of their lumbar spine will be analyzed in detail from CT and MRI imaging (morphological measurements of their vertebra and the intervertebral discs). Another one-hundred and fifty CT and MRI imaging of non symptomatic low back group will be taken from the "Meir medical center" in order to characterize the symptomatic group and their degenerative changes.

ELIGIBILITY:
Inclusion Criteria:

* Participants' diagnosis may include unstable degenerative spondylolisthesis, radicular pain, or documented stenosis with referred pain

Exclusion Criteria:

* Psychiatric illness
* Previous spine surgery
* Painful arthritic hip
* Hospitalization or surgery in the previous 6 months
* Alcohol consumption > 10 drinks/week
* Diabetes or other causes for poly neuropathy
* Metabolic bone disease, tumor, spinal deformity or contraindications to MRI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CLBP (>12 weeks) and degenerative changes of the lumbar spine confirmed by CT imaging who were recommended surgery and chose to undergo surgery will be recruited from the department of Orthopedic Surgery at the Meir Medical Center, Kfar-Saba, and in Assuta hospital, Tel Aviv, Israel. Included participants will be men or women, aged 40-80 years, of any race or ethnic background. Participants' diagnosis may include unstable degenerative spondylolisthesis, radicular pain, or documented stenosis with referred pain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06-15 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change in Oswestry Disability Index (ODI) score which is equal to or greater than 50% has been used consistently in Physical Therapy literature as the definition of success following an intervention | 6 weeks pre-op, 1 month post op, 6 months post op and 1 year post op
The Roland Morris Disability Questionnaire (RMQ) | up to 1 year
  Commonly used in CLBP research as measures of patients' participation restrictions

SECONDARY OUTCOMES:
The Fear Avoidance Beliefs questionnaire (FABQ) | 6 weeks pre-op, 1 month post op, 6 months post op and 1 year post op
  The FABQ was found to be an important prognostic factor for work-related outcomes in patients with sub-acute LBP and a component of clinical predictors rules predicting changes in ODI following physical therapy interventions for patients with LBP
The International Physical Activity Questionnaire (IPAQ) | 6 weeks pre-op, 1 month post op, 6 months post op and 1 year post op
  The IPAQ was designed to provide a set of well-developed instruments that can be used internationally to obtain comparable estimates of physical activity
The Visual Analog Scale (VAS) | 6 weeks pre-op, 1 month post op, 6 months post op and 1 year post op
  The VAS is one of the most commonly used pain measures in CLBP research and has been shown to be reliable in this population
Lumbar myotomes function | 6 weeks pre-op, 6 months post op and 1 year post op
  Will be taken by the Hand-held dynamometry (HHD) in order to assess the lower extremity muscle force output
The Long Distance Corridor Walk (LDCW) | 6 weeks pre-op, 6 months post op and 1 year
  comprised of a 2 minute warm up and a 400 meter walk as fast as possible
The 8 foot up and go | 6 weeks pre-op, 6 months post op and 1 year
  The 8-foot version of the Time-up-and-go test is part of the reliable and valid senior fitness test. Performance on the test indicates on sensory, motor, strength and balance function
The 30-seconds chair stand test | 6 weeks pre-op, 6 months post op and 1 year
  for lower body strength
Grip strength | 6 weeks pre-op, 6 months post op and 1 year
  Hand grip strength was found to be associated with changes in disability and pain following aquatic therapy in patients with CLBP
single leg stance test | 6 weeks pre-op, 6 months post op and 1 year
  measures static balance
The four square step test | 6 weeks pre-op, 6 months post op and 1 year
  measures dynamic balance
Passive straight leg raise (PSLR) | 6 weeks pre-op, 6 months post op and 1 year
  Passive straight leg raise (PSLR) up to first sensation of pain will be measured with an inclinometer

OTHER OUTCOMES:
Morphological parameters | 6 weeks pre-op
  morphological parameters in the lumbar spine will be analyzed from the CT imaging : a) Lumbar lordosis b) Sacral angle orientation, c) Pelvic tilt , d) Pelvis width e) Lumbar vertebral body and disc shape- the vertebral body and inter-vertebral disc lengths, widths, heights and wedging ,Lumbar vertebral arch shape

CONTACTS AND LOCATIONS:
Overall Officials: Youssef Masharawi, DPT, Study Chair — Tel Aviv University
Locations (1):
- Assuta hospital, Tel Aviv, Israel

REFERENCES:
- [Background] Maniadakis N, Gray A. The economic burden of back pain in the UK. Pain. 2000 Jan;84(1):95-103. doi: 10.1016/S0304-3959(99)00187-6. PMID 10601677
- [Background] Dankaerts W, O'Sullivan PB, Burnett AF, Straker LM. The use of a mechanism-based classification system to evaluate and direct management of a patient with non-specific chronic low back pain and motor control impairment--a case report. Man Ther. 2007 May;12(2):181-91. doi: 10.1016/j.math.2006.05.004. Epub 2006 Jul 31. No abstract available. PMID 16877024
- [Background] Matsui H, Maeda A, Tsuji H, Naruse Y. Risk indicators of low back pain among workers in Japan. Association of familial and physical factors with low back pain. Spine (Phila Pa 1976). 1997 Jun 1;22(11):1242-7; discussion 1248. doi: 10.1097/00007632-199706010-00014. PMID 9201863
- [Background] Lundon K, Bolton K. Structure and function of the lumbar intervertebral disk in health, aging, and pathologic conditions. J Orthop Sports Phys Ther. 2001 Jun;31(6):291-303; discussion 304-6. doi: 10.2519/jospt.2001.31.6.291. PMID 11411624
- [Background] Masharawi YM, Peleg S, Albert HB, Dar G, Steingberg N, Medlej B, Abbas J, Salame K, Mirovski Y, Peled N, Hershkovitz I. Facet asymmetry in normal vertebral growth: characterization and etiologic theory of scoliosis. Spine (Phila Pa 1976). 2008 Apr 15;33(8):898-902. doi: 10.1097/BRS.0b013e31816b1f83. PMID 18404110
- [Background] Luoma K, Riihimaki H, Luukkonen R, Raininko R, Viikari-Juntura E, Lamminen A. Low back pain in relation to lumbar disc degeneration. Spine (Phila Pa 1976). 2000 Feb 15;25(4):487-92. doi: 10.1097/00007632-200002150-00016. PMID 10707396
- [Background] Ammendolia C, Chow N. Clinical outcomes for neurogenic claudication using a multimodal program for lumbar spinal stenosis: a retrospective study. J Manipulative Physiol Ther. 2015 Mar-Apr;38(3):188-94. doi: 10.1016/j.jmpt.2014.12.006. Epub 2015 Jan 22. PMID 25620608
- [Background] Delitto A, Erhard RE, Bowling RW. A treatment-based classification approach to low back syndrome: identifying and staging patients for conservative treatment. Phys Ther. 1995 Jun;75(6):470-85; discussion 485-9. doi: 10.1093/ptj/75.6.470. PMID 7770494
- [Background] Lubetzky-Vilnai A, Ciol M, McCoy SW. Statistical analysis of clinical prediction rules for rehabilitation interventions: current state of the literature. Arch Phys Med Rehabil. 2014 Jan;95(1):188-96. doi: 10.1016/j.apmr.2013.08.242. Epub 2013 Sep 10. PMID 24036159
- [Background] Abbas J, Hamoud K, May H, Hay O, Medlej B, Masharawi Y, Peled N, Hershkovitz I. Degenerative lumbar spinal stenosis and lumbar spine configuration. Eur Spine J. 2010 Nov;19(11):1865-73. doi: 10.1007/s00586-010-1516-5. Epub 2010 Jul 21. PMID 20652366
- [Background] Singh K, Samartzis D, Vaccaro AR, Nassr A, Andersson GB, Yoon ST, Phillips FM, Goldberg EJ, An HS. Congenital lumbar spinal stenosis: a prospective, control-matched, cohort radiographic analysis. Spine J. 2005 Nov-Dec;5(6):615-22. doi: 10.1016/j.spinee.2005.05.385. PMID 16291100